CLINICAL TRIAL: NCT04532203
Title: Clinical Trial for the Safety and Efficacy of CAR-T Cells Therapy for Patients With the Central Nervous System Involvement of Relapsed and/or Refractory B-cell Acute Lymphoblastic Leukemia or B-cell Non-Hodgkin's Lymphoma
Brief Title: A Study of CAR-T Cells Therapy for Patients With Relapsed and/or Refractory Central Nervous System Hematological Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNSL-ZhejiangU
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma
Keywords: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; CAR T-cell therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CAR T-cells (Experimental): Dose escalation follows the standard 3+3 doseescalation design. A total of 3 dose levels are set for subjects.
  Interventions: Drug: CAR-T cells; Procedure: Ommaya Reservoir

INTERVENTIONS:
Drug: CAR-T cells — Each subject receive CAR T-cells by intravenous infusion
  Other Names: CAR-T cells injection
Procedure: Ommaya Reservoir — Surgical catheter placement into the fourth ventricle of the brain

SUMMARY:
A Study of CAR-T Cells Therapy for Patients With Relapsed and/or Refractory Central Nervous System Hematological Malignancies

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory central nervous system CD19+ B-cell hematological malignancies, including acute lymphoblastic leukemia and B-cell non-Hodgkin's lymphoma. The selections of dose levels and the numberof subjects are based on clinical trialsof similar foreign products. Two groups of patients will be enrolled, 36 in eachgroup. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria only for B-ALL:

  1. Male or female aged 3-70 years;
  2. Histologically confirmed diagnosis of B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
  3. Relapsed or refractory CD19+ B-ALL (meeting one of the followingconditions):

     1. CR not achieved after standardized chemotherapy;
     2. CR achieved following the first induction, but CR duration isless than 12 months;
     3. Ineffectively after first or multiple remedial treatments;
     4. 2 or more relapses;
  4. The number of primordial cells (lymphoblast and prolymphocyte)in bone marrow is>5% (by morphology), and/or >1% (by flowcytometry);
  5. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphia-chromosome-positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;
* Inclusion criteria only for B-NHL:

  1. Male or female aged 18-75 years;
  2. Histologically confirmed diagnosis of DLBCL (NOS), FL, DLBCL transformed from CLL/SLL, PMBCL, and HGBCL per the WHOClassification Criteria for Lymphoma (2016);
  3. Relapsed or refractory B-NHL (meeting one of the followingconditions):

     1. No response or relapse after second-line or abovechemotherapy regimens;
     2. Primary drug resistance;
     3. Relapse after auto-HSCT;
  4. At least one assessable tumor lesion per Lugano 2014 criteria;
* Common inclusion criteria for B-ALL and B-NHL:

  1. Highly suspected or confirmed central nervous system involvement of hematological malignancies;
  2. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit ofnormal, creatinine ≤ 176.8 umol/L;
  3. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
  4. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
  5. Estimated survival time ≥ 3 months;
  6. ECOG performance status 0 to 2;
  7. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance,epilepsy,cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinarytractinfectionand bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving inhaled steroids;
7. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts,orbilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk ofpatients or interfere with the results of study.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell acute lymphocytic leukemia(B-ALL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
B-ALL, Overall survival (OS) | Up to 2 years after CAR-T cells infusion
  From the first infusion of CAR-T cells to death or the last visit
B-ALL, Event-free survival (EFS) | Up to 2 years after CAR-T cells infusion
  From the first infusion of CAR-T cells to the occurrence of any event, including death, relapse orgene relapse, disease progression (any one occurs first), and the last visit
B cell non-hodgkin's lymphoma (B-NHL), Overall response rate (ORR) | At Week 4, 12, and Month 6, 12, 18, 24
  Assessment of ORR (ORR = CR + PR) per Lugano 2014 criteria
B-NHL, disease control rate (DCR) | At Week 12 and Month 6, 12, 18, 24
  Assessment of DCR (DCR=CR+PR+SD) per Lugano 2014 criteria
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Quality of life using Research and Treatment of Cancer QOL Core Questionnaire 30 (EORTC QLQ-30) at Baseline, Month 1, 3, 6, 9 and 12
IADL score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of IADL score at Baseline, Month 1, 3, 6, 9 and 12
ADL score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of ADL score at Baseline, Month 1, 3, 6, 9 and 12
HADS score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Hospital Anxiety and Depression Scale (HADS) score at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No